CLINICAL TRIAL: NCT03788083
Title: A Phase I Study on the Safety and Immune-modulatory Effect of Intratumoral (i.t.) Administration of mRNA (Messenger RNA) Encoding Dendritic Cell Activating Proteins in Patients With Early, Resectable Breast Cancer
Brief Title: Intratumoral TriMix Injections in Early Breast Cancer Patients
Acronym: TMBA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: eTheRNA immunotherapies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TriMix-Breast
Record Dates: First submitted 2018-11-16; First posted 2018-12-27 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer Female; Early-stage Breast Cancer
Keywords: immune therapy; dendritic cells; immune priming
MeSH Terms: conditions — Breast Neoplasms | interventions — trimix

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects will not know whether an active or non-active substance is being injected. The choice for TriMix or placebo will take place according to the predefined schedule and can not be influenced by the patient or the investigator. Only after the comparison of the tumour tissue before (the initial biopsy where the diagnosis was made) and after (obtained at second biopsy or surgery) the intratumoral injection, it will be known whether mRNA or non-active product was used for the injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- TriMix (Active Comparator)
  Interventions: Drug: Trimix

INTERVENTIONS:
Drug: Trimix — Intratumoral TriMix injection
  Arms: TriMix
Drug: Placebo — Intratumoral placebo injection
  Arms: placebo

SUMMARY:
Patients with early breast cancer and accessible tumor lesions (1.00 to 10 ml volume) that are eligible to either surgical removal of their tumor or neoadjuvant chemotherapy will be injected with the IMP. Patients will be either treated with placebo (buffer alone, 12 patients) or with TriMix mRNA at three dose levels [8 at dose level I (1mg/ml), 8 at dose level II (3mg/ml), and 8 at dose level III (6mg/ml). The volume injected in this group will be adjusted to the tumour volume to ensure a perfusion of around 33% of the tumour volume (33% +/- 5%). Therefore, depending on the patients' tumour size, 500, 1000 or 2000 µl of TriMix mRNA solution or placebo solution will be injected into each tumor. Each patient will receive three administrations of TriMix prior to start of general treatment (surgery or neoadjuvant chemotherapy) separated by one week (7 days +/- 2 days) interval. The last administration will be performed 2 days preoperatively or start of neoadjuvant chemotherapy.

The tumor and peripheral blood samples will be analyzed for immunological changes. If it is decided by the multidisciplinary team that neoadjuvant therapy is more appropriate for the patient, a second tumor biopsy (instead of surgical resection) will be taken 2 days after third administration of TriMix mRNA to assess immunological changes within the tumor. Similarly, patients that refuses to undergo surgery or to receive neoadjuvant chemotherapy can be enrolled into the trial, if they accept three administrations of TriMix followed by a second tumor biopsy.

The study will start with recruitment of the placebo group. The enrollment of the first three patients in each cohort with Trimix mRNA will be staggered with at least one day between the first dose of each individual patient. One week after the third patient of a cohort received the third TriMix mRNA administration, an overall evaluation of the safety and tolerability of this cohort will be done by the principal investigator. The results will be reviewed by an in-house dose evaluation committee overseeing the safety and tolerability of TriMix mRNA.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years and less than or equal to 85 yrs
2. Histologically proven breast cancer eligible for curative surgery (with or without the need for neoadjuvant chemotherapy) with one or more injection-accessible (allowing ultrasound guidance) nodal tumors.
3. Injectable tumor lesions must have a volume between 1.00 and 10 ml, only one lesion per patient will be injected
4. ECOG performance status of 0 or 1
5. Willing to give informed consent in writing
6. Willing and able to attend the scheduled study visits and to comply with the study procedures
7. No prior therapy for ipsilateral breast cancer
8. Normal lab parameters: white cell count ≥ 3,000/mm3, hemoglobin ≥ 10mg/dl, platelet count ≥ 100,000/mm3, serum creatinine ≤ 1.5 x institutional ULN, bilirubin ≤ 2.0 mg/dl aspartate aminotransferase/alanine aminotransferase/ alkaline phosphatase ≤ 2 x the upper normal limit (AST< 72 U/l, ALT < 104 U/l, AP < 252 U/l)
9. Adequate Coagulation Parameters with: Prothrombin INR < 1.5; Partial Thromboplastin Time < 1.5 x 34.4 sec (51.6 sec)
10. Female patients of childbearing potential should have a negative serum pregnancy test at screening visit and should use a highly efficient method of birth control for the duration of treatment and until the first menses after a 4 week period after the last dose of study medication. Highly effective birth control methods include:

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation administered oral, intravaginal or transdermal.
    * progestogen-only hormonal contraception associated with inhibition of ovulation administered oral, as an injectable or implantable formulation.
    * intrauterine device
    * intrauterine hormone-releasing system
    * bilateral tubal occlusion
    * vasectomised partner
    * abstinence from sexual intercourse

Exclusion Criteria:

1. Male patients
2. Patients with stage III-IV breast cancer (AJCC 8th edition)
3. Patients with highly vascularized tumor or important post-biopsy hematoma
4. Previous chemotherapy for breast cancer or other types of cancer within the last five years
5. Other malignancies other than non-melanoma skin cancer, or controlled superficial bladder cancer. In the event of prior malignancies treated surgically, the patient must be considered NED (no evidence of disease) for a minimum of 3 years prior to enrolment
6. Patients with a history of autoimmune disease (inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, rheumatoid arthritis or multiple sclerosis) other auto-immune or debilitating diseases. Vitiligo is not an exclusion criterion.
7. Patients with serious intercurrent chronic or acute illness such as pulmonary [asthma or chronic obstructive pulmonary disease (COPD)] or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the P.I. to constitute an unwarranted high risk for investigational drug treatment
8. Patients with significant psychiatric disabilities or seizure disorders
9. Legal incapacity or limited legal capacity
10. Patients on steroid therapy > 10 mg prednisone (or equivalent) or other immunosuppressive agents such as azathioprine or cyclosporine A are excluded on the basis of potential immune suppression. Patients must have had 8 weeks of discontinuation of any steroid therapy exceeding > 10 mg prednisone (or equivalent) prior to enrolment
11. Presence of an active acute or chronic infection, including symptomatic urinary tract infection, HIV (as determined by ELISA and confirmed by Western Blot) or viral hepatitis (as determined by HBsAg and Hepatitis C serology)
12. Patient is pregnant or is currently breast-feeding

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 2 years
  Number of patients with adverse events, total number of adverse events, dose limiting toxicities

SECONDARY OUTCOMES:
Tumor microenvironment changes induced by intratumoral TriMix mRNA | 30 days
  Tumor microenvironment changes induced by intratumoral TriMix mRNA administration from diagnostic biopsy to day 21 (visit 5) assessed by immunohistochemistry.
Tumor microenvironment changes induced by intratumoral TriMix mRNA | 30 days
  Tumor microenvironment changes induced by intratumoral TriMix mRNA administration from diagnostic biopsy to day 21 (visit 5) assessed by nanoString gene profiling
TriMix mRNA induced T-cell responses | 30 days
  TriMix mRNA induced T-cell responses assessed by immunoassays in situ and in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Marian Vanhoeij, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium